CLINICAL TRIAL: NCT04942574
Title: Voice Biomarkers to Predict Excessive Daytime Sleepiness
Acronym: SOMVOICE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Bordeaux (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: CHUBX 2020/57
Record Dates: First submitted 2021-06-18; First posted 2021-06-28 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Sleep Deprivation
Keywords: Sleep Deprivation; Voice biomarkers; sleepiness
MeSH Terms: conditions — Sleep Deprivation; Sleepiness

STUDY DESIGN:
Intervention Model Description: This is a monocentric exploratory study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- First experimental visit : Total Sleep Deprivation (Experimental): The participants enrolled in this arm will have a total sleep deprivation on their first experimental visit and a normal sleep on their second experimental visit.
  Interventions: Other: Total sleep deprivation; Other: Normal sleep
- First experimental visit : Normal Sleep (Experimental): The participants enrolled in this arm will have a normal on their first experimental visit and a total sleep deprivation sleep on their second experimental visit.
  Interventions: Other: Total sleep deprivation; Other: Normal sleep

INTERVENTIONS:
Other: Total sleep deprivation — Participants will perform repeatedly : task of reading with voice acquisition before each MSLT, KSS, VAS-Anxiety, VAS-Fatigue and PVT during the day after a night of total sleep deprivation.
Other: Normal sleep — Participants will perform repeatedly : task of reading with voice acquisition before each MSLT, KSS, VAS-Anxiety, VAS-Fatigue and PVT during the day after a night of normal sleep.

SUMMARY:
This study aims at measuring the impact of a night of sleep deprivation over the vocal characteristics of healthy subjects.To do so, the subjects takes a Multiple Sleep Latency Test (MSLT) the day after a night of total sleep deprivation (or a supervised normal night for the control subjects). Before each iteration of the MSLT, the subjects are recorded during the reading of a text and fill three medical questionnaires : Karolinska Sleepiness Scale (KSS), Visual Analogue Scale for Fatigue (VAS-F) and Visual Analogue Scale for Anxiety (VAS-A), allowing to link variations of vocal markers to the variations of these measures.

DETAILED DESCRIPTION:
Excessive Daytime Sleepiness (EDS) is a frequent symptom that concerns between 5% and 8% of the population. The individual consequence of EDS is a diminution of the life quality. Furthermore, EDS is a cause of high socio-medical costs though the accidental risks that it induces at work and on the road (Ohayon, Reynolds et al. 2013). Indeed, it is a severe symptom due to the consequences that it is the cause of. Furthermore, EDS is associated to 5 to 20% of road accidents depending on the type of road network. As a consequence, to elaborate a sleepiness detection through voice in real time system is a major challenge for public health-care and medicine. Moreover, it offers benefits from a socio-medical aspect, as detecting sleepiness through voice doesn't require neither consumables furniture nor specialized staff to be set up.

To highlight the effect of sleepiness over voice, investigators designed this experiment around a night of total sleep deprivation. To measure objective sleepiness of subjects, they takes a MSLT test the day after a night of total sleep deprivation (or a supervised night for control). The complementary measures (KSS, VAS-A, VAS-F and Psychomotor Vigilance Task (PVT)) will allow to study the exact origin of the variations of the vocal markers induced by the sleep deprivation.

ELIGIBILITY:
Inclusion Criteria:

* Male ou female volunteers, who are between 18 and 50 years old,
* With a BMI (Body Mass Index) between 18.5 and 25 kg/m2 for volunteers who are between 18 and 34 years old, or a BMI between 18.5 and 27 kg/m2 for volunteers who are between 35 and 50 years old ,
* Not having subjective EDS (Excessive Daytime Sleepiness) : total score at ESS (Epworth Sleepiness Scale) lower or equal to 11,
* Not having insomnia complaints (ISI total score lower than 8),
* Having a SCL90R (Symptom Check List- 90 items Revised) score lower than 60 (only for Anxiety and Depression categories' items of the checklist),
* Regular bedtime between 22H00 and 0H00, regular get up time between 6H00 and 8H00,
* Daily TST (Total Sleep Time) between 7 and 9 hours,
* With no strong suspicion of OSAS (Obstructive Sleep Apnea Syndrome) as assessed by STOP-BANG questionnaire,
* With no suspicion of RLS (Restless Legs Syndrome) as assessed by RLS screening questionnaire,
* With sufficient reading abilities for the reading task as assessed by ECLA16+ ("Evaluation des Compétences de Lecture chez l'Adulte de plus de 16 ans" :

higher ou equal performances than 25th percentile for performances assessed in total population for the following tasks : " lecture de " l'Alouette " " (Number of correctly read words / minute ≥ 121, number of errors ≤ 10), isolated words reading (regular words : score ≥ 18, time ≤ 17 sec ; irregular words : score ≥ 16, time ≤ 16 sec, pseudo-words : score ≥ 17, time ≤ 26 sec), repetition of non-words (score ≥ 19), and symbol crossing task (number of crossed symbols ≥ 22),

* With a SE (Sleep Efficiency) higher or equal to 85% as assessed by the 7 nights-actigraphy made before inclusion,
* With an AHI (Apnea/Hypopnea Index) lower or equal to 10 apnea or hypopnea/hour of sleep as assessed by the ventilatory polygraphy,
* With a PLMI (Periodic Limb Movement Index) lower or equal to 15 sequences of PLM/hour of sleep as assessed by the ventilatory polygraphy,
* Being an affiliated member of the Social Security system,
* Being able to understand the study,
* Being available to come at the four visits necessary for the study,
* Having given written informed consent to participate to the study.

Exclusion Criteria:

* Having a life-threatening disease,
* Any evolutive cardiovascular pathology - under treatment or not,
* Any evolutive neurologic pathology - under treatment or not (brain tumour, epilepsy, headache, stroke, sclerosis, myoclonia, chorea, neuropathy, muscular dystrophies, myotonic dystrophy),
* Psychiatric disorders - under treatment or not (characterised depressive episode, bipolar disorders, psychotic disorders, neurodevelopmental diseases),
* Untreated endocrine disorders (diabetes, hyperthyroidism),
* Dependency to a substance,
* otorhinolaryngological disorder that could induce vocal parameters modification,
* Fluence disorders (cluttering, stuttering), language disorders (dyslexia) or visual troubles that could impact reading abilities,
* Participant under psychotropic treatment (antidepressants, antihistamine, etc…), or under treatment that could interfere with sleep or wakefulness level,
* Participant under treatment that could impact the normal muscular function (myorelaxant, neuromuscular blocking agents injections in maxillofacial area, etc…),
* Dental care during the follow-up of the study,
* Shift-worker or night-worker,
* Excessive consumption of alcohol (>2 glasses per day) during the 6 last months,
* Excessive consumption of coffee, tea, or any drink containing caffeine (like cola) (> 5 cups/day),
* Excessive tobacco smoking (>5 cigarets/day),
* Non-native French speaker,
* Participant with a thick accent that could induce significantly vocal parameters modification (at the discretion of the investigator),
* Deprived of liberty by a legal or administrative procedure,
* Under tutorship or guardianship,
* Pregnant or breastfeeding woman.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2022-02-07 (Actual); Primary Completion 2024-06-10 (Actual); Study Completion 2024-06-10 (Actual)

PRIMARY OUTCOMES:
Acoustic fingerprint | Visit 3 (V3) between 14 and 60 days after inclusion (V1)
  Acoustic fingerprint (statistics on prosody, frequency and energy) influenced by sleep deprivation measured at each iteration of TILE at visits V2 and V3.

SECONDARY OUTCOMES:
sleep onset | Visit (V2) between 7 and 10 days after inclusion (V1) and Visit 3 (V3) between 14 and 60 days after inclusion (V1)
  The sleep onset at each iteration of the MSLT (in minutes). This evaluate the objective sleepiness of the subject, right after that its voice has been recorded, allowing to link vocal markers and objective sleepiness of the subject.
Karoslinska Sleepiness Scale questionnaire | Visit (V2) between 7 and 10 days after inclusion (V1) and Visit 3 (V3) between 14 and 60 days after inclusion (V1)
  The score to the Karoslinska Sleepiness Scale questionnaire. This measure links the vocal markers with subjective instantaneous sleepiness.
  Minimum value 1 (extremely alert); maximum value 9 (extremely sleepy, fighting sleep)
VAS-Fatigue | Visit (V2) between 7 and 10 days after inclusion (V1) and Visit 3 (V3) between 14 and 60 days after inclusion (V1)
  The score to the VAS-Fatigue. This measure links the vocal markers and with the fatigue of the subject.
  Visual analog scale from minimum (energetic, no fatigue) to maximum (worst fatigue possible)
VAS-Anxiety. | Visit (V2) between 7 and 10 days after inclusion (V1) and Visit 3 (V3) between 14 and 60 days after inclusion (V1)
  The score to the VAS-Anxiety. This measure links the vocal markers and the anxiety level of the subject.
  Visual analog scale from minimum (calm) to maximum (anxious)
PVT | Visit (V2) between 7 and 10 days after inclusion (V1) and Visit 3 (V3) between 14 and 60 days after inclusion (V1)
  The score to the PVT . This links the vocal markers of the subject to its level of performance.
lexical decision | Visit (V2) between 7 and 10 days after inclusion (V1) and Visit 3 (V3) between 14 and 60 days after inclusion (V1)
  The scores to the lexical decision task

CONTACTS AND LOCATIONS:
Locations (1):
- CHU de Bordeaux, Bordeaux, France

IPD SHARING:
Plan to Share IPD: No